CLINICAL TRIAL: NCT00216983
Title: Proline Metabolism in Severely Burned Patients: Effect of Modulated Parenteral Feeding.
Status: Withdrawn | Type: Observational
Why Stopped: State of Mass. tightened regulations for making intravenous solutions for research subjects. Study was withdrawn and no participants were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ronald G. Tompkins, MD, ScD, Chief, Burn Service, Massachusetts General Hospital
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Other Study IDs: 1999-P-008463; 2P50GM021700-27 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Burns
Keywords: parenteral nutrition; burn injury; stable isotopes; Proline Metabolic Kinetics; Ornithine Metabolic Kinetics; Glutamate Metabolic Kinetics; Glutamine Metabolic Kinetics
MeSH Terms: conditions — Burns; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Fasting condition to measure:
  1. quantitative relationships among proline, ornithine and glutamate with an emphasis on evaluating the rate of proline disposal and its conversion to ornithine and glutamate in burn patients
  2. Evaluating the rate of proline de novo synthesis from glutamate or ornithine in burn patients
- 2: We will study the quantitative relationships among proline, ornithine and glutamate with an emphasis on evaluating the rate of proline disposal and its conversion to ornithine and glutamate in burn patients. When the patients are receiving regular TPN or TPN depleted with proline - arginine - glutamate.
- 3: We wull evaluate the rate of proline de novo synthesis from glutamate or ornithine in burn patients when the patients are receiving regular TPN or TPN depleted proline-arginine-glutamate.

SUMMARY:
The overall purpose of the study is to evaluate the effect of depleting proline supply in the nutritional support regimen on proline metabolism in the burn patients, this includes the rate of proline oxidation after burn injury, the rate of proline de novo synthesis from its immediate precursors glutamate and ornithine. The specific aims of the proposed study are: 1) to determine the kinetic status of proline metabolism and whole body proline balance under the following nutritional states: (a) "fasting; (b) regular total parenteral nutrition (TPN); (c)TPN with isonitrogenous depletion of proline, glutamate and ornithine metabolism under nutritional conditions studied in specific aim 1) above.

DETAILED DESCRIPTION:
Proline is a non-essential amino acid. Its synthesis and catabolism is via the pathway of ornithine and glutamate, the latter two amino acids serve as its immediate precursors as well as metabolites. Ornithine is one of the intermediates for urea cycle, and glutamate is metabolically connected to tricarboxylic acid (TCA) cycle, the major cycle for energy production.

It is hypothesized that the significantly increased rates of net nitrogen loss and energy "production", as the consequence of the accelerated activities of both the urea and TCA cycles in burn injury "drain" both ornithine and glutamate, thus depleting tissues of the availability of proline. Hence, the de novo synthesis of proline is likely to be affected by the reduced availability of its major precursors: glutamate and ornithine.

This hypothesis is supported by 1) tissue and circulating glutamine content are reduced in stressed conditions; 2) ornithine disposal via oxidation is significantly increased after burn injury(2). Therefore, the availability of proline is likely to be limiting after burn injury for the synthesis of proteins. On the other hand, proline requirement is significantly increased in burn patients due to the high demand for tissue repair and wound healing. As a result, providing an adequate proportion of its precursors, glutamine / glutamate and / or as preformed proline, is of importance to maintain the appropriate supply and balance of amino acids for protein and other synthetic functions after burn injury.

The overall purpose of the study is to evaluate the effect of depleting proline supply in the nutritional support regimen on proline metabolism in the burn patients, this includes the rate of proline oxidation after burn injury, the rate of proline de novo synthesis from its immediate precursors glutamate and ornithine. The specific aims of the proposed study are: 1) to determine the kinetic status of proline metabolism and whole body proline balance under the following nutritional states: (a) "fasting; (b) regular total parenteral nutrition (TPN); (c)TPN with isonitrogenous depletion of proline, glutamate and ornithine metabolism under nutritional conditions studied in specific aim 1) above.

ELIGIBILITY:
Inclusion Criteria:

Burn patients being treated at MGH Burn Unit with one or more of the following criteria: 1) >=5% TBSA; 2) inhalation injury; or 3) resting energy expenditure (REE) of >15% of the predicted Basal Metabolic Rate using the Harris-Benedict equation.

Must be receiving total parenteral nutrition in the course of their treatment.

Exclusion Criteria:

Patients with thyroid disease. Patients who are not hemodynamically stable or show unstable vital signs Patients at the stage of major organ failure, e.g. renal and/or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill burn patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1997-09; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
This is a study for measuring the protein kinetics for metabolism of the amino acid proline kinetics will be derived from measurements on blood and air samples taken as part of the study. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital - Boston
Locations (1):
- Massachusetts General Hospital Burn Unit, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tharakan JF, Yu YM, Zurakowski D, Roth RM, Young VR, Castillo L. Adaptation to a long term (4 weeks) arginine- and precursor (glutamate, proline and aspartate)-free diet. Clin Nutr. 2008 Aug;27(4):513-22. doi: 10.1016/j.clnu.2008.04.014. Epub 2008 Jun 30. PMID 18590940
- [Background] Yu YM, Ryan CM, Castillo L, Lu XM, Beaumier L, Tompkins RG, Young VR. Arginine and ornithine kinetics in severely burned patients: increased rate of arginine disposal. Am J Physiol Endocrinol Metab. 2001 Mar;280(3):E509-17. doi: 10.1152/ajpendo.2001.280.3.E509. PMID 11171607
- [Background] Yu YM, Ryan CM, Burke JF, Tompkins RG, Young VR. Relations among arginine, citrulline, ornithine, and leucine kinetics in adult burn patients. Am J Clin Nutr. 1995 Nov;62(5):960-8. doi: 10.1093/ajcn/62.5.960. PMID 7572742
- [Background] Jaksic T, Wagner DA, Burke JF, Young VR. Proline metabolism in adult male burned patients and healthy control subjects. Am J Clin Nutr. 1991 Aug;54(2):408-13. doi: 10.1093/ajcn/54.2.408. PMID 1858705
- [Background] Jaksic T, Wagner DA, Burke JF, Young VR. Plasma proline kinetics and the regulation of proline synthesis in man. Metabolism. 1987 Nov;36(11):1040-6. doi: 10.1016/0026-0495(87)90023-0. PMID 3670073